CLINICAL TRIAL: NCT04343690
Title: Effectiveness of Crisis Management Coaching on Faculty and Trainee Wellness During COVID-19 Crisis
Brief Title: COPING With COVID-19( CWC-19)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Ended May 1, 2020 with no enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00105319
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Care Workers (Experimental): Faculty, staff, and trainees dealing with COVID-19 pandemic
  Interventions: Behavioral: Crisis management coaching

INTERVENTIONS:
Behavioral: Crisis management coaching — Crisis management coaching will be offered to faculty, staff, and trainees dealing with COVID-19 pandemic

SUMMARY:
The purpose of this study is 1) to understand effects of COVID-19 crisis on wellness of pulmonary and critical care faculty and trainees who are at frontline fighting this pandemic 2) Assess the effectiveness of series of weekly web based crisis management coaching from world renowned experts in coaching and 3) identify future areas of opportunities in physician wellness

ELIGIBILITY:
Inclusion Criteria:

* Any faculty, staff, or trainee from Duke pulmonary and critical care that consents to being in the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in stress level as measured by survey | Baseline, mid-session (up to 4 weeks), post-intervention (up to 8 weeks)

SECONDARY OUTCOMES:
Change wellness as measured by survey | Baseline, mid-session (up to 4 weeks), post-intervention (up to 8 weeks)
  Survey is 14-items asking about wellness on a scale from "Strongly Agree" to "Not at all"

CONTACTS AND LOCATIONS:
Overall Officials: Patty Lee, MD, Principal Investigator — Duke University; Sangeeta Joshi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No